CLINICAL TRIAL: NCT06069518
Title: Continuous Glucose Monitoring as a Strategy to Optimize Metabolic Control in Patients With Diabetes on Peritoneal Dialysis Therapy Entitled to the IMSS
Brief Title: Continuous Glucose Monitoring in Patients With Diabetes on Peritoneal Dialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: R-2023-785-072; R-2023-785-072 (Other Grant/Funding Number: Baxter Healthcare Corporation)
Record Dates: First submitted 2023-10-02; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Kidney Disease, Chronic; Peritoneal Dialysis; Diabetes Mellitus Type 2
Keywords: remote monitoring; Continuous glucose monitoring; peritoneal dialysis; diabetes mellitus; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: The patient presenting Chronic Kidney Disease, with etiology of diabetes mellitus (DM), has a metabolic alteration characterized by an elevation of glycemia and accompanied by cardiovascular complications, this increases the morbidity and mortality associated with the disease. Therefore, it is necessary to maintain adequate metabolic control to reduce the incidence of these complications. This task is extraordinarily difficult without the use of Icodextrin due to the optimal adjustment of insulin, due to the additional supply of glucose contained in the Dialysis Bosas and which is absorbed through the peritoneum.

Under this premise, it is of utmost importance the surveillance of the patient through constant glycemic monitoring to provide an overview of the metabolic status of our patients, this will allow clinically relevant data to improve care, minimize expenses in the health system and implement measures for decision making in the adjustment of dialysis treatment.

Objective: To use continuous glucose monitoring to detect whether the type, dose, route of administration and timing of insulin application are associated with the patterns provided by continuous glucose monitoring (magnitude and duration of periods of hyper and/or hypoglycemia) in 24-hour periods of tissue glucose.

Material and methods: This is a cross-sectional, non-interventional study in adult patients with Type 2 Diabetes Mellitus on Peritoneal Dialysis in its Automated modality who present high and high average peritoneal transport type.

As inclusion criteria, participants over 40 years of age, of any sex, diagnosed with Diabetic Nephropathy, and who are insulin-dependent for metabolic control, with at least three months of PD treatment. The project will consist of evaluating the patient's glycemic control continuously, with an automatic scan and data recording every six hours during the infusion time of Automated Peritoneal Dialysis. For this, 110 patients are required according to the sample size. The Guardian TM 3 Sensor will be placed using the One PressTM Grafter subcutaneously in the upper posterior region of the patient's non-dominant arm, it is a minimally invasive procedure that does not require surgical protocols. This sensor will be connected to the Guardian Connect Transmitter for continuous communication with the Guardian™ Connect (App).

The sensor has an approximate life of 7 days (time that lasts the enzymatic reaction and that allows an adequate measurement) the data will be transmitted every five minutes 24 hours a day, for 7 consecutive days. The patient will be scheduled at the end of these days to place a second sensor and complete the 14 days of follow-up.

On day seven, the patient will be scheduled for sensor removal, and a new one will be placed to complete 14 days of follow-up. On day 14, the total 24-hour PD drainage volume will be recovered for a glucose, urea and creatinine measurement and peritoneal glucose absorption, D/P creatinine and Kt/V will be calculated. The dietary information will be obtained for the calculation of calorie intake and meal time; it is together with the subcutaneous application of insulin will be recorded within the same GuardianTM Connect (App).

Statistical analysis: The databases will be audited in monthly periods by random sampling in blocks of 5% of their content. Semi-annual reports will be integrated with the monitoring of the records achieved and the outcomes to date of the reports. The reports will contain the basic descriptive information (central tendency and dispersion) according to the characteristics of the variables. Patients will be classified according to the time of glucose measurements within the pre-established ranges (70-180 mg / dL), the goal is that 70% of the time they are in that range and will be called "Adequate" and those who do not reach the goal will be called "Not Adequate".

The results will be reported with measures of central tendency and dispersion appropriate to the characteristics of the variables. For the detection of difference between the appropriate and inappropriate group, the Chi square statistic or the Student's T or Mann-Whitney U will be used according to the type of variables.

For the association analysis that allows detecting the variables of greatest influence on glycemic control in the recommended ranges with continuous glucose monitoring, logistic regression analysis will be used. In a first stage, analysis will be done by independent variable and in a second stage, a multivariate analysis will be made, where the type of insulin, the route of administration, the dose and the schedules will be considered. At this stage, confounding variables will also be included, such as; obesity, adherence to treatment and diet and physical activity prescribed by the treating physician.

DETAILED DESCRIPTION:
JUSTIFICATION The high prevalence of patients with end-stage CKD treated with PD and the dominant frequency of DM as a cause of CKD make it necessary to have documented guidelines for the metabolic control of patients with DM who use PD.

Guidelines should consider the use of insulin in terms of dose, which should be consistent with the supply of glucose in food and the amount absorbed from the peritoneum. Consistent also with the meal schedule and infusion schedules of PD solutions with higher glucose concentration, as well as with the route of administration, since the peritoneal route requires up to twice the dose applied subcutaneously.

To generate these guidelines, monitoring metabolic control with conventional tools, such as serum glucose concentrations with portable glucometer or glycosylated hemoglobin, is inoperative because they do not allow identifying the times of day when insulin should be applied to optimize its use. Continuous glucose monitoring is the only practical tool available that can be used for this purpose.

In recent reports, CKD stands out as the 3rd chronic-degenerative disease with the greatest financial impact for the IMSS, which together with diabetes mellitus and hypertension consume most of the total care expenditure of chronic patients. Moreover, patients with DM are more than half of patients on dialysis programs.

With the panorama described, it is evident that metabolic control and water balance in patients with DM on PD becomes both a clinical and economic challenge.

RESEARCH QUESTION Is continuous glucose monitoring an effective tool to detect the effect of the type, dose, route of administration and timing of insulin on metabolic control in patients with diabetes and on peritoneal dialysis? OBJECTIVES General Objective Use continuous glucose monitoring to detect whether the type, dose, route of administration, and timing of insulin application are associated with the patterns provided by continuous glucose monitoring (magnitude and duration of periods of hyper- and/or hypoglycemia) in 24-hour periods of tissue glucose.

Specific Objectives To identify the patterns of insulin prescription in patients with diabetes on PD (type, dose, schedule of application, route of administration).

Compare the daily profile of glucose concentration measured by continuous monitoring with the fasting glucose concentration and with the percentage of glycosylated hemoglobin.

Detect which insulin administration scheme is associated with shorter times and magnitude of hypo and hyperglycemia.

Measure the peritoneal absorption of glucose and its parallelism with glucose measured by continuous monitoring.

MATERIAL AND METHODS Design: Cross-sectional study without intervention. Population: Adult patients with type 2 diabetes mellitus (DM2) with terminal CKD being treated with peritoneal dialysis.

Inclusion criteria: Participants over 40 years of age, of any sex, diagnosed with Diabetic Nephropathy, and who are exclusively insulin-dependent for metabolic control, with at least three months of PD treatment.

Non-inclusion criteria: Patients with positive serology for HIV and hepatitis B and C, acute complications and hospitalization for cardiovascular, metabolic or infectious disease in the month prior to inclusion in the study, cancer, pregnancy or allergy.

Outcomes Primary: Average glucose concentration detected in 24-hour periods. Magnitude and duration of periods1s of hiccups (<70 mg/dl) and hyperglycemia (>180 mg/dl) recorded in 24-hour periods.

Secondary: Necessary adjustments in insulin dose during the surveillance period.

Procedures Patients who meet the admission criteria (in the PD consultation records) will be invited to participate in the study by a member of the research group. They will be informed of the objective of the study and the procedures involved.

From patients who agree to participate and have signed the informed consent letter, the first interview will collect demographic data (gender, age, marital status, education, economic activity, income) clinical (original disease, time of evolution, previous hospitalizations, comorbidity) and laboratory (blood biometrics, basic biochemistry of inflammation, mineral metabolism, nutrition and cardiovascular) contained in their file. The information will be collected by nursing staff trained in the development of Clinical Research projects (Monitors). The data to be collected are those established as dialysis adequacy criteria and are specified in the attached formats.

They will be cited for the collection of blood samples that will serve for the biochemical analysis that includes: glucose, urea, creatinine, total cholesterol, HDL cholesterol, triglycerides, glycosylated hemoglobin and C-reactive protein.

They will be trained in the management of the glucose monitor which will be placed in the non-dominant arm. Once the monitor is calibrated, the patient will be monitored for seven days, after which the sensor will be removed and another sensor will be placed to have a sum of fourteen days of follow-up.

The recorded data will be collected by the researchers and kept in sheets designed for that purpose.

The training of patients is of theoretical-practical face-to-face type in which, it will be verified that they do the procedures of calibration and consultation of their glucose properly and that they understand the meaning of the prevention signals so that they have security in the use of the monitor.

If glucose concentrations above 250 mg / dL are recorded in a timely manner or periods of more than 7 hours (30%) per day, the patient will be sent to a detailed review by his treating physician, who will be previously warned of the metabolic lack of control.

Laboratory. All biochemical and laboratory tests will be used for routine surveillance of the patient on PD and will be performed at the Hospital of affiliation with usual automated techniques.

Continuous Glucose Monitoring. GuardianTM 3 sensor. Guardian Connect Transmitter Kit and Guardian Connect System, consisting of Guardian Connect Transmitter, One PressMT Grafter and Guardian™™™TM Connect Smartphone App (App), Generic printing equipment Said sensor will be connected to the Guardian™ Connect Transmitter for continuous communication with the GuardianTM Connect (App). For this, it is necessary to have a Smartphone, in case of not having said telephone device, one will be given to the patient so that they can carry out the follow-up properly.

After a proven proper functioning, through the calibration supported by the use of a Glucometer and reactive strips for capillary glycemia, the data will be transmitted every five minutes, 24 hours a day, for 7 consecutive days (time that the enzymatic reaction lasts and that allows an adequate measurement) the patient will be summoned at the end of these days to place a second sensor and complete the 14 days of follow-up.

The information provided by the GuardianTM Connect system is downloadable in Excel format, and can also be analyzed by the clinician from the CareLinkTM website. Trends, patterns in glucose concentration and main alerts outside the established range will be analyzed.

On day 7, the patient will be called to remove the sensor and the total 24-hour PD drainage volume will be recovered for a measurement of glucose, urea, and creatinine. Likewise, peritoneal glucose absorption, D/P creatinine will be calculated. and Kt/V. Diet information will be obtained to calculate calorie intake and meal time, along with the subcutaneous application of insulin will be recorded within the same GuardianTM Connect (App).

Statistical plan The databases will be audited in monthly periods by random sampling in blocks of 5% of their content.

Semi-annual reports will be integrated with the monitoring of the records achieved and the outcomes up to the date of the reports. The reports will contain the basic descriptive information (central tendency and dispersion) according to the characteristics of the variables.

Patients will be classified according to the time of glucose measurements within the pre-established ranges (70-180 mg/dL) (24), the goal is that 70% of the time they are in that range and will be called "Adequate" and those that do not reach the goal will be called "Not Adequate".

The results will be reported with measures of central tendency and dispersion appropriate to the characteristics of the variables.

To detect the difference between the adequate and non-adequate groups, the Chi-square statistic or the Student's T or Mann-Whitney U test will be used according to the type of variables.

For the association analysis that allows the detection of the variables with the greatest influence on glycemic control in the recommended ranges with continuous glucose monitoring, logistic regression analysis will be used. In the first stage, an analysis will be carried out by independent variable, and in the second stage, a multivariate analysis will be carried out, where the type of insulin, the route of administration, the dose, and the schedules will be considered. In this stage, the confounding variables will also be included, such as; obesity, adherence to treatment, and diet and physical activity prescribed by the treating physician.

By protocol, the independent variables considered will be daily glucose absorption, insulin dose, application time with respect to food intake and PD solutions used, as well as the route of administration. All the analyzes will be carried out with the statistical program SPSS v24. The significance level will be p<0.05.

Sample size

The following assumptions were used to calculate the sample size:

Statistical test to apply: Logistic regression. Dependent variable: Time of tissue glucose concentration in range (dichotomized as "Adequate" or "Not Adequate") Dominant covariate: Insulin administration route (dichotomized as ("Subcutaneous" or "Intraperitoneal"). It is considered the most important covariate because it is the one associated with better control in studies where punctual glucose concentration was used as an indicator of metabolic control. with a portable glucometer and/or glycosylated hemoglobin.

α: 0.05 β: 0.9 OR: Risk of time out of range >85%: (Intraperitoneal/Subcutaneous) 0.46/0.30. N: 110 Ethical aspects

The research will be governed by the ethical principles and guidelines stipulated in the Official Mexican Standard NOM-028-SSA2-1999 and the General Health Law on research in human beings according to articles 96 and 100 of Title V and the Technical Standard number 313. These laws confer the degree of protection of the person in relation to respect for their rights, dignity, well-being, and anonymity. The guidelines to be followed will be the following:

An informed consent letter is included, which will be presented to the patient by associated researchers who are duly accredited before the authorities of the participating Medical Units.

In accordance with the Regulations of the General Health Law on Health Research 1984, Articles 21, where it is stated: For informed consent to be considered existing, the research subject or, where appropriate, their legal representative You must receive a clear and complete explanation, in such a way that you can understand it, at least, on the following aspects.

This research is considered to be of minimal risk since it involves common procedures in physical examinations for routine diagnoses or treatments, coupled with the use of a proven device with evidence in the literature that will provide new parameters for the metabolic control of patients with diabetes. The use of this device does not imply risk since its placement is intradermal, it does not imply risk of venous bleeding or direct application of insulin. The alarms that it potentially generates will be detected by the patient, who will previously be instructed in their meaning and what he must do. According to clinical experience in the control of patients with PD, the observed glucose variations are within ranges that do not imply a risk for the patient but that allow for optimizing the application of insulin.

If glucose concentrations exceeding 250 mg/dL are recorded in a timely manner or for periods of more than 7 hours (30%) a day, the patient will be sent for a detailed review by his treating physician, who will be previously warned of metabolic uncontrolled.

The risk/benefit balance is positive since, with minimal risk, the potential value of the information is relevant.

It should be noted that none of the participating researchers have any conflict of interest with the use of the GuardianTM Connect device.

The samples will be handled by experienced personnel and prepared at each center since only glycosylated hemoglobin and clinical laboratories will be taken prior to the patient's monthly consultation.

For this, it is declared that the General Health Law in Research Matters and the regulations and biosafety manuals are known and have been read, for which the following points are cited.

Regarding installing the Guardian Connect Sensor, there is training for the personnel that will install it. For installation, there is training provided by the "Latam Medtronic Academy" to minimize risks, and control and manage its installation material.

No sample will be processed within the laboratory since the pieces from it will be processed in each center to avoid the transfer of serum or blood plasma. It is also highly recommended to use adequate personal protective equipment when installing the sensor on patients on dialysis.

Resources, financing, and feasibility The research team is made up of a nephrologist with experience in the hospital patient clinic, a nephrology area researcher, and two nurses, in addition, there is an electronic capture of information by trained personnel to do so.

The expected surplus costs derive from the need to have electronic devices for glycemic monitoring, which will be requested resources for the development of this.

The research group has proven experience in various publications in the nephrology context.

ELIGIBILITY:
Inclusion Criteria: Participants over 40 years of age, of any sex, diagnosed with Diabetic Nephropathy, and who are exclusively insulin-dependent for metabolic control, with at least three months of PD treatment.

Exclusion Criteria: Patients with positive serology for HIV and hepatitis B and C, acute complications, and hospitalization for cardiovascular, metabolic or infectious disease in the month prior to inclusion in the study, cancer, pregnancy, or allergy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the admission criteria (in the PD consultation records) will be invited to participate in the study by a member of the research group. They will be informed of the objective of the study and the procedures involved.
  From patients who agree to participate and have signed the informed consent letter, the first interview will collect demographic data (gender, age, marital status, education, economic activity, income) clinical (original disease, time of evolution, previous hospitalizations, comorbidity) and laboratory (blood biometrics, basic biochemistry of inflammation, mineral metabolism, nutrition and cardiovascular) contained in their file. The information will be collected by nursing staff trained in the development of Clinical Research projects (Monitors). The data to be collected are those established as dialysis adequacy criteria and are specified in the attached formats.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Average glucose concentration detected in 24-hour periods. | 14 days of follow-up
  Amount of time that blood glucose is within the target range during and after dialysis fluid infusion. Measurement of time in which blood glucose levels are within the lower range of 70 mg/dL and an upper range of 180 mg/dL during and after the infusion of dialysis fluid.

SECONDARY OUTCOMES:
Magnitude and duration of periods1s of hiccups (<70 mg/dl) and hyperglycemia (>180 mg/dl) recorded in 24-hour periods. | 14 days of follow-up
  Presence of hypoglycemia (glucose concentration less than 70 mg/dL) or hyperglycemia (glucose concentration greater than 180 mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: José Ramón Paniagua Sierra. R Paniagua,, PhD, Study Director — Unidad de Investigación Médica en Enfermedades Nefrológicas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ng JKC, Ling J, Luk AOY, Lau ESH, Ma RCW, Li PKT, Szeto CC, Chan JCN, Chow E. Evaluation of a Fourth-Generation Subcutaneous Real-Time Continuous Glucose Monitor (CGM) in Individuals With Diabetes on Peritoneal Dialysis. Diabetes Care. 2023 Jun 1;46(6):1191-1195. doi: 10.2337/dc22-2348. PMID 37043824
- [Background] Bomholt T, Kofod D, Norgaard K, Rossing P, Feldt-Rasmussen B, Hornum M. Can the Use of Continuous Glucose Monitoring Improve Glycemic Control in Patients with Type 1 and 2 Diabetes Receiving Dialysis? Nephron. 2023;147(2):91-96. doi: 10.1159/000525676. Epub 2022 Jul 13. PMID 35830847
- [Background] Almalki MH, Altuwaijri MA, Almehthel MS, Sirrs SM, Singh RS. Subcutaneous versus intraperitoneal insulin for patients with diabetes mellitus on continuous ambulatory peritoneal dialysis: meta-analysis of non-randomized clinical trials. Clin Invest Med. 2012 Jun 1;35(3):E132-43. doi: 10.25011/cim.v35i3.16589. PMID 22673316
- [Background] Galindo RJ, Beck RW, Scioscia MF, Umpierrez GE, Tuttle KR. Glycemic Monitoring and Management in Advanced Chronic Kidney Disease. Endocr Rev. 2020 Oct 1;41(5):756-74. doi: 10.1210/endrev/bnaa017. PMID 32455432
- [Background] Selby NM, Fonseca S, Hulme L, Fluck RJ, Taal MW, McIntyre CW. Hypertonic glucose-based peritoneal dialysate is associated with higher blood pressure and adverse haemodynamics as compared with icodextrin. Nephrol Dial Transplant. 2005 Sep;20(9):1848-53. doi: 10.1093/ndt/gfh946. Epub 2005 Jun 21. PMID 15972319